CLINICAL TRIAL: NCT00961961
Title: Prevention of Relapse & Recurrence of Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH080097 (NIH); R01MH080097 (NIH); R01MH080098 (NIH)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Manic Depression; Major Depressive Episode; Mania; Hypomania; Long Term Treatment
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Lithium; Fluoxetine; Lithium Carbonate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lithium plus Fluoxetine Phase I (Other): All participants were started in this arm. Those who met criteria for entry into Phase II were then randomized to one of the two Phase II arms.
  Interventions: Drug: Lithium / Fluoxetine
- Lithium plus Placebo Phase I (Other): No participants began their participation on Lithium plus Placebo.
  Interventions: Drug: Lithium / Placebo
- Lithium plus Fluoxetine Phase II (Experimental): Patients who responded to Lithium plus Fluoxetine in Phase I and were randomized to continue on both compounds.
  Interventions: Drug: Lithium / Fluoxetine
- Lithium plus Placebo Phase II (Placebo Comparator): Patients who responded to Lithium plus Fluoxetine in Phase I and were randomized to switch from Fluoxetine to placebo.
  Interventions: Drug: Lithium / Placebo

INTERVENTIONS:
Drug: Lithium / Fluoxetine — Individualized Daily Dosage
  Other Names: Lithium Carbonate / Prozac
  Arms: Lithium plus Fluoxetine Phase I; Lithium plus Fluoxetine Phase II
Drug: Lithium / Placebo — Individualized Daily Dosage
  Other Names: Lithium Carbonate / Sugar Pill
  Arms: Lithium plus Placebo Phase I; Lithium plus Placebo Phase II

SUMMARY:
The purpose of this study is to determine whether the long-term use of combined antidepressant plus mood stabilizer therapy is superior to mood stabilizer therapy alone in preventing the relapse and recurrence of bipolar depression.

DETAILED DESCRIPTION:
Recurrence of Bipolar I (BP I) major depressive episode (MDE), is now recognized as a major mental health problem. Recurrent BP I MDE is a disorder with no satisfactory therapy, and its treatment remains a challenge to clinicians. To date, initial and long-term therapy of BP I MDE has been based on un-validated practice guidelines. These guidelines recommend limiting antidepressant drug (AD) use during initial therapy of BP I MDE, and completely avoiding AD use during long-term therapy. There is, however, no empirical evidence to suggest that mood stabilizer (MS) monotherapy is superior to combined MS plus AD therapy in preventing recurrent BP I MDE. Nor is there evidence to suggest that long-term MS plus AD therapy results in more manic switch episodes. We present evidence that AD-induced mania during long-term therapy of BP I MDE has been over-estimated, and that long-term use of MS plus AD therapy may be superior to MS therapy alone in preventing recurrent BP I MDE. In this study, we will ask: "Does continuation therapy with combined lithium plus fluoxetine result in fewer MDE relapses and recurrences vs. lithium monotherapy?" To answer this question, patients with BP I MDE will receive combined lithium plus fluoxetine therapy for 8 weeks. Responders who stay well for an additional 4 weeks of consolidation therapy will then be randomized to double-blind continuation therapy with either (i) combined lithium plus fluoxetine, or (ii) lithium alone (following fluoxetine taper and discontinuation) for an additional 50 weeks. We hypothesize that long-term lithium plus fluoxetine therapy will result in fewer MDE relapses and recurrences vs. lithium monotherapy. We will also ask: "What is the relative safety, tolerability, and frequency of syndromal and sub-syndromal manic, hypomanic, and mixed state conversions during continuation treatment with combined lithium plus fluoxetine vs. lithium monotherapy?" To answer this question, we will measure: the frequency, severity, and duration of syndromal and sub-syndromal manic, hypomanic, and mixed state conversions; frequency, severity, and duration of treatment-emergent adverse events; frequency of treatment discontinuation; time to onset of first syndromal and sub-syndromal conversion event; time to first treatment intervention of each syndromal and sub-syndromal conversion event; and, time to onset of increase in suicidal ideation event. We hypothesize that lithium plus fluoxetine therapy will result in a similar frequency of syndromal and sub-syndromal conversion events, and a similar frequency of treatment-emergent adverse events. We further hypothesize that lithium plus fluoxetine therapy will result in fewer suicide ideation events and fewer study discontinuations vs. lithium monotherapy. We believe that the results of this trial may have an important public health impact on the current practice guidelines for treating BP I MDE.

ELIGIBILITY:
Inclusion Criteria:

* Men/women (all races and ethnicity)
* Age at least 18 years old
* Bipolar Type I Disorder
* Current Major Depressive Episode
* Able to understand and provide signed informed consent

Exclusion Criteria:

* Current alcohol or drug abuse
* Alcohol or drug dependence within 3 months
* Allergic to Fluoxetine or Lithium
* Unstable medical condition (e.g., uncontrolled thyroid, renal, cardiovascular disease)
* Pregnant or nursing women
* Women of child-bearing potential unwilling to use a medically acceptable form of contraception
* Actively suicidal
* Requiring hospitalization
* Use of medication contraindicated with lithium or fluoxetine
* Unable to participate in a year-long trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. DeRubeis, PhD, Principal Investigator — University of Pennsylvania; John M Zajecka, MD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Depression Research Unit, Philadelphia, Pennsylvania

REFERENCES:
- See also: DeRubeis Lab Web Page — http://web.sas.upenn.edu/derubeis/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I was an open label treatment, of Lithium and Fluoxetine, of all enrolled patients.
  Those who met criteria for response after 12 weeks were randomized to one of two Phase II (double-blinded) arms:
  Lithium plus Fluoxetine
  Lithium plus Placebo
Groups:
- Lithium Plus Placebo Phase I: This is a placeholder arm. No participants were given Placebo in Phase I.
- Lithium Plus Fluoxetine Phase II: One of the two randomly assigned groups, each of which continued on Lithium Double-blind assignment to continue on Fluoxetine (this group)
- Lithium Plus Placebo Phase II: One of the two randomly assigned groups, each of which continued on Lithium Double-blind assignment to switch from Fluoxetine to Placebo (this group)
Period: Phase I
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
Started | 177 | 0 | 0 | 0
Completed | 51 | 0 | 0 | 0
Not Completed | 126 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0 | 0
Not completed — Lack of Efficacy | 94 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0 | 0
Not completed — Physician Decision | 8 | 0 | 0 | 0
Period: Phase II
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
Started | 0 (This is a Phase I category. Not relevant in Phase II.) | 0 (This is a Phase I category. Not relevant in Phase II.) | 29 | 22
Completed | 0 | 0 | 17 | 14
Not Completed | 0 | 0 | 12 | 8
Not completed — Lost to Follow-up | 0 | 0 | 10 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants were assessed prior to entering the open label phase of the study.
Groups:
- Lithium Plus Fluoxetine Phase I: All eligible and consenting participants began in this open phase. Therefore baseline characteristics are only relevant for this category.
- Lithium Plus Placebo Phase I: No participant was begun on Placebo. Lithium Plus Placebo was a real condition only after randomization, in Phase II. Baseline characteristics for all participants are listed under Lithium plus Fluoxetine Phase I.
- Lithium Plus Fluoxetine Phase II; Lithium Plus Placebo Phase II: This is a subset of patients whose baseline characteristics are listed under Lithium plus Fluoxetine Phase I.
- Total: Total of all reporting groups
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II | Total
Number analyzed (Participants) | 177 | 0 | 0 | 0 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 175 | 0 | 0 | 0 | 175
  >=65 years | 2 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 0 | 0 | 0 | 90
  Male | 87 | 0 | 0 | 0 | 87
Region of Enrollment [Number; unit: participants]
  United States | 177 |  |  |  | 177

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse of Major Depressive Episode Within 1 Year
Description: Patients who were randomized to one of the Phase II conditions were interviewed once each month. If they met criteria for a relapse of a Major Depressive Episode, this was considered the study outcome. If they participated for the full year of Phase II without a documented relapse, they were considered a completer.
Time Frame: 1 year
Population: The analyses are relevant only during Phase II. The comparisons are between those assigned to one of the two randomized Phase II conditions.
Measure: Count of Participants; unit: Participants
Groups:
- Lithium Plus Fluoxetine Phase I; Lithium Plus Placebo Phase I: The outcome measures, including this one, are only relevant in Phase II. Thus there will be zeroes in this category.
- Lithium Plus Fluoxetine Phase II: Participants randomized to this condition remained on active medications. However, the fluoxetine pills were made to look like the placebo pills, to maintain the double-blind.
- Lithium Plus Placebo Phase II: Participants randomized to this condition were switched from fluoxetine to placebo. However, the placebo pills were made to look like the fluoxetine pills, to maintain the double-blind.
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
Number analyzed (Participants) | 0 | 0 | 29 | 22
Participants |  |  | 4 | 5

2. Secondary Outcome: Number of Participants With an Onset of a Manic Episode Within 1 Year
Description: Onsets of a manic episodes were ascertained with the clinician-rated Young Mania Rating Scale (YMRS). The YMRS covers 11 symptom groups over the previous 48 hours. Four of the items are rated on a scale from 0 to 4; the other 4 are rated on a scale of 0 to 8. A score of 12 or above indicates a manic episode.
Time Frame: 1 Year
Population: This and other outcomes are only relevant in the double-blind Phase II of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Lithium Plus Fluoxetine Phase I; Lithium Plus Placebo Phase I: This is not a relevant category for this outcome. This outcome is only assessed in Phase II.
- Lithium Plus Fluoxetine Phase II: Includes participants who completed Phase I and were assigned randomly to continue on their medications in Phase II (double-blind, as the fluoxetine and placebo were identical in appearance.
- Lithium Plus Placebo Phase II: Includes participants who completed Phase I and were assigned randomly to switch from fluoxetine to placebo in Phase II (double-blind, as the fluoxetine and placebo were identical in appearance).
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
Number analyzed (Participants) | 0 | 0 | 29 | 22
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With an Onset of a Hypomanic Episode Within 1 Year
Description: Onsets of a hypomanic episodes were ascertained with the clinician-rated Hypomania Interview Guide and associated scoring rules.
Time Frame: 1 Year
Population: These are the patients who were randomly assigned, after responding to the medications provided in Phase I, to either remain on the same regime or have their fluoxetine switched to placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Lithium Plus Fluoxetine Phase I: All participants began with both medications in Phase I, which led into Phase II.
- Lithium Plus Placebo Phase I: No participant was on placebo in Phase I. Only during Phase II.
- Lithium Plus Placebo Phase II: Participants randomized to this condition were switched from fluoxetine to placebo. However, the fluoxetine pills were made to look like the placebo pills, to maintain the double-blind.
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
Number analyzed (Participants) | 0 | 0 | 29 | 22
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With the Onset of a Sub-Syndromal Mood Conversion Episode Within 1 Year
Time Frame: 1 Year
Population: This was not a diagnosis that was recognized widely in the profession. Procedures for ascertaining such episodes were not consistent across the two performance sites. As a consequence the data obtained to document this outcome were unreliable.
Groups:
- Lithium Plus Fluoxetine: Lithium / Fluoxetine: Individualized Daily Dosage
- Lithium Plus Placebo: Lithium / Placebo: Individualized Daily Dosage
- Lithium Plus Placebo Phase II: Participants randomized to this condition remained on active medications. However, the fluoxetine pills were made to look like the placebo pills, to maintain the double-blind.
Arm/Group | Lithium Plus Fluoxetine | Lithium Plus Placebo | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 15 months
Description: All events were noted during the first phase of the study.
Groups:
- Lithium Plus Fluoxetine Phase I: This is the condition that all participants started in. They were given Lithium plus Fluoxetine and, if they responded, they were asked to accept random assignment to Phase II.
- Lithium Plus Placebo Phase I: No one was on placebo in Phase I.
- Lithium Plus Fluoxetine Phase II: These are the patients randomly assigned to stay on the fluoxetine in Phase II.
- Lithium Plus Placebo Phase II: These are the patients randomly assigned to switch to placebo from fluoxetine in Phase II.
Arm/Group | Lithium Plus Fluoxetine Phase I | Lithium Plus Placebo Phase I | Lithium Plus Fluoxetine Phase II | Lithium Plus Placebo Phase II
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/0 | 0/29 | 0/22
Serious Adverse Events (participants affected / at risk) | 20/177 | 0/0 | 0/29 | 0/22
Other Adverse Events (participants affected / at risk) | 0/177 | 0/0 | 0/29 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Plus Fluoxetine Phase I (N=177) | Lithium Plus Placebo Phase I (N=0) | Lithium Plus Fluoxetine Phase II (N=29) | Lithium Plus Placebo Phase II (N=22)
Suicide ideation (Psychiatric disorders) | 2 (2) | NA | 0 | 0
Acute mood disturbance (Psychiatric disorders) | 2 (2) | NA | 0 | 0
Elevated Creatinine (Gastrointestinal disorders) | 1 (1) | NA | 0 | 0
Unable to swallow pills (Gastrointestinal disorders) | 1 (1) | NA | 0 | 0
Hospitalized for dehydration (General disorders) | 1 (1) | NA | 0 | 0
Hospitalized for overdose of benzodiazepines (Psychiatric disorders) | 2 (2) | NA | 0 | 0
Hospitalized for acute alcohol abuse (Psychiatric disorders) | 1 (1) | NA | 0 | 0
Hospitalized for acute substance abuse (Psychiatric disorders) | 1 (2) | NA | 0 | 0
Lethargy, cognitive dulling (Nervous system disorders) | 3 (3) | NA | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | NA | 0 | 0
Muscle stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | 0 | 0
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | NA | 0 | 0
Tremors (Nervous system disorders) | 3 (3) | NA | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No